CLINICAL TRIAL: NCT05641077
Title: Are Virtual Visits for Delivery of Postoperative Care Following Urogynecologic Surgery Equal to Office Visits? The VIDEO Randomized Trial
Brief Title: Virtual Visits for Postoperative Care Following Urogynecologic Surgery
Acronym: VIDEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-1269
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-06

CONDITIONS: Satisfaction, Patient
Keywords: Urogynecology; Virtual visit; Telehealth; Urogynecologic surgery; Healthcare resource utilization; Patient satisfaction; Postoperative
MeSH Terms: conditions — Patient Satisfaction | interventions — Office Visits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Visit (Experimental): Patients randomized to the experimental arm will be scheduled for and follow up with the surgeon or an advanced practice provider via a virtual visit using videoconference technology at 6 weeks after the anticipated date of surgery. If the surgery were to be rescheduled to a future date, the postoperative visit will be moved accordingly to ensure follow-up occurs at the 6-week postoperative period.
  Interventions: Other: Virtual Visit
- Office Visit (Active Comparator): Patients randomized to the active comparator arm will be scheduled for and follow up with the surgeon or an advanced practice provider via an in-office visit at 6 weeks after the planned date of surgery. If the surgery were to be rescheduled to a future date, the postoperative visit will be moved accordingly to ensure follow-up occurs at the 6-week postoperative period.
  Interventions: Other: Office Visit

INTERVENTIONS:
Other: Virtual Visit — Patients randomized to this arm will be scheduled for and follow up with the surgeon or an advanced practice provider via a virtual visit using videoconference technology at 6 weeks after the anticipated date of surgery. If the surgery were to be rescheduled to a future date, the postoperative visit will be moved accordingly to ensure follow-up occurs at the 6-week postoperative period.
  Arms: Virtual Visit
Other: Office Visit — Patients randomized to this arm will be scheduled for and follow up with the surgeon or an advanced practice provider via an in-office visit at 6 weeks after the planned date of surgery. If the surgery were to be rescheduled to a future date, the postoperative visit will be moved accordingly to ensure follow-up occurs at the 6-week postoperative period.
  Arms: Office Visit

SUMMARY:
The proposed VIDEO randomized trial will help inform clinical practice regarding the utility and perceived value of videoconferencing for postoperative care of urogynecologic patients by comparing patient satisfaction with virtual video visits and traditional in-office visits after pelvic organ prolapse and/or anti-incontinence surgery. Patient satisfaction will be measured by the Patient Satisfaction Questionnaire-18 at the 6-week postoperative visit. The investigators hypothesize that patient satisfaction with the virtual postoperative visit will be non-inferior to an in-office visit. The study will secondarily investigate other important components of healthcare quality, including safety and clinical outcomes, by comparing postoperative healthcare resource utilization and adverse events within 12 weeks after urogynecologic surgery. Healthcare resource utilization as measured by patient-initiated phone calls, unscheduled in-person/virtual office visits, emergency room or urgent care visits, and inpatient readmissions within 6 weeks following surgery and within 12 weeks following surgery. The study also aims to evaluate patient and provider preferences/attitudes toward in-office versus virtual-video postoperative visits.

DETAILED DESCRIPTION:
The study is a randomized controlled noninferiority trial evaluating patient satisfaction with in-office versus virtual-video postoperative visits at six weeks following urogynecologic surgery. We aim to assess whether the intervention of virtual postoperative visit via videoconference technology is noninferior to the standard/traditional in-office postoperative visit for our primary outcome of patient satisfaction. The recruitment period will be 15 months (January 1, 2023 to March 31, 2024). The follow-up period for each participant will be 12 weeks after surgery.

The investigators will recruit patients of the Center for Urogynecology and Pelvic Reconstructive Surgery in the Department of Obstetrics/Gynecology and Women's Health Institute at the Cleveland Clinic scheduled to undergo major or minor surgery for pelvic organ prolapse and/or urinary incontinence. Participants will be prospectively identified by the primary surgeon during the patient's initial consultation when the decision is made to proceed with surgery for pelvic organ prolapse and/or urinary incontinence. Enrolled participants will be randomized to either the office visit arm or the virtual visit arm. Stratified block randomization will be used to ensure that the number of participants is equally distributed among the study groups and stratified by surgery level (major, minor).

Study instruments will be administered at the preoperative visit and the 6-week postoperative visit. The questionnaires for this study include the Patient Preparedness Questionnaire (PPQ), the Patient Satisfaction Questionnaire-18 (PSQ-18), and modified patient and provider preference questionnaires entitled, Patient Postoperative Visit Questionnaire and Provider Postoperative Visit Preference Questionnaire.

In addition to questionnaire responses, the investigators will collect the following information from the electronic medical record: Demographic data (e.g. age, race, parity, body mass index), perioperative data (e.g. surgery level major/minor, surgery type, concomitant procedures, estimated blood loss, operative time), six-week postoperative data (e.g. route of postoperative visit in-office/virtual, patient-initiated phone calls to surgeon's office, unanticipated outpatient visits, emergency department visits, hospital readmissions prior to the postoperative visit, adverse events prior to postoperative visit), and 6-12 week postoperative data (e.g. patient-initiated phone calls to surgeon's office, unanticipated outpatient visits, emergency department visits, hospital readmissions, and adverse events after the scheduled postoperative visit for up to 12 weeks after surgery).

A priori sample size calculation determined that 100 participants (50 per group) would allow for 80% power to assess a noninferiority margin of 5 points on the total PSQ-18, with a SD of 10 and significance level of 0.05. A minimum important difference has not been reported for the PSQ-18; however, previous studies using this tool demonstrated SD for total PSQ-18 score ranging between 2.6 and 11.8 and used a 5-point interval for the noninferiority margin. To account for an anticipated attrition rate of approximately 5%, we aimed to enroll a total of 106 participants (53 per group).

Patient satisfaction (PSQ-18) total scores, as well scores in each of the 7 PSQ-18 domains, will be treated as continuous data and checked for normality. Healthcare utilization will be analyzed individually (number of phone calls, number of outpatient visits, number of emergency department or urgent care visits, number of hospital readmissions), as well as a composite of all encounter types. Adverse events will be analyzed independently but also as a composite utilizing the Clavien-Dindo Grading System for surgical complications. Attitudes toward office/virtual visits will be analyzed by comparing proportions of patients and providers who prefer a virtual visit, prefer an office visit, or have no preference.

All analyses will be conducted using an intention-to-treat principle. Baseline demographic and clinical characteristics will be summarized using descriptive statistics. Normally-distributed continuous measures will be summarized using mean and standard deviation (SD), whereas those showing departure from normality will be summarized using median and interquartile range (IQR). Categorical measures will be summarized using number of participants and percentage. The primary end-point analysis will be designed to test whether patient satisfaction with a virtual postoperative visit is noninferior to an in-person postoperative visit, as determined by the total PSQ-18 at the scheduled postoperative visit. Noninferiority would be shown if the lower limit of the two-sided 95% confidence interval for the between-group mean difference in the primary endpoint (i.e., the difference between the mean PSQ-18 total score in the virtual group minus the mean PSQ-18 total score in the in-office group) is more than -5 points. Similar analyses will be performed for each secondary outcome. The noninferiority margin is defined as 5 points for the PSQ-18 total score and 0.5 points for the PSQ-18 domain scores, 10% absolute for composite healthcare resource utilization, and 25% absolute for composite adverse events. Planned exploratory subgroup analyses of patient satisfaction, healthcare resource utilization and adverse events based on surgery level will be additionally performed. All statistical analyses will be performed using JMP Pro version 17.0 software (SAS Institute, Cary, NC). Data will be managed in REDCap. Statistical support will be provided by the Cleveland Clinic Quantitative Health Sciences.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* Has technological capability to participate in videoconferencing (high-speed internet access with desktop computer or mobile device)
* Has decision-making capacity and able to provide informed consent for research participation
* Able to speak and read English

Exclusion Criteria:

* Patient requested to physically come in the office or have a virtual visit for her postoperative visit
* Planned concomitant surgery with another surgical team
* Office follow-up is deemed medically necessary by provider/surgeon

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Urogynecological post-operative study
Enrollment: 100 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile A Ferrando, M.D., M.P.H., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Lua-Mailland LL, Nowacki AS, Paraiso MFR, Park AJ, Wallace SL, Ferrando CA. Virtual Compared With In-Office Postoperative Visits After Urogynecologic Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2024 Oct 1;144(4):562-572. doi: 10.1097/AOG.0000000000005694. Epub 2024 Aug 8. PMID 39116443

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Visit | Office Visit
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Visit | Office Visit | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 35 | 64
  >=65 years | 21 | 15 | 36
Age, Continuous [Mean (Full Range); unit: Years] | 58.4 [28 to 80] | 55.5 [31 to 77] | 57 [28 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 44 | 47 | 91
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: Patient satisfaction will be measured by the Patient Satisfaction Questionnaire-18 (PSQ-18) at the 6-week postoperative visit. The PSQ-18 is a validated 18-item questionnaire. Responses to each question are scored on a five-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). The total score for the questionnaire ranges from 18 (dissatisfaction with medical care) to 90 (highest satisfaction with medical care).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Visit | Office Visit
Number analyzed (Participants) | 50 | 50
score on a scale | 75.18 (8.15) | 75.14 (8.7)

ADVERSE EVENTS:
Time Frame: Participants were followed for up to 12 weeks after surgery.
Arm/Group | Virtual Visit | Office Visit
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT05641077/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT05641077/ICF_001.pdf